CLINICAL TRIAL: NCT00233259
Title: CHD Lifestyle Modification for Latinas With Diabetes
Brief Title: Lifestyle Modification Program to Reduce Risk of Coronary Heart Disease in Latina Women With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 327; R01HL076151 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2 | interventions — Diet, Mediterranean; Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Multiple risk factor intervention, that will include diet, physical activity, stress management, social support, and smoking cessation components
  Interventions: Behavioral: Mediterranean Diet; Behavioral: Physical Activity; Behavioral: Stress Management; Behavioral: Social Support; Behavioral: Smoking Cessation
- 2 (Placebo Comparator): Control group
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Mediterranean Diet — Mediterranean dietary program
  Arms: 1
Behavioral: Physical Activity — Physical activity program
  Arms: 1
Behavioral: Stress Management — Stress management program
  Arms: 1
Behavioral: Social Support — Social support
  Arms: 1
Behavioral: Smoking Cessation — Smoking cessation program
  Arms: 1
Other: Control group — Usual Diabetes Care Control group
  Arms: 2

SUMMARY:
The Viva Bien! trial will comprehensively evaluate a multiple risk factor intervention (diet, physical activity, stress management, social support, and smoking cessation) in a randomized effectiveness trial, which will be offered in English and Spanish to diabetic Latinas.

DETAILED DESCRIPTION:
BACKGROUND:

Age-adjusted mortality from coronary heart disease (CHD) has been increasing in women with diabetes. On the other hand, it has been decreasing in women without diabetes and in men with and without diabetes. CHD remains the leading cause of death among women in the United States. Risks of CHD and resulting death are significantly higher among postmenopausal women; these rates are two and a half times higher among women with diabetes versus women without diabetes. Diabetes is an independent risk factor for CHD in both Latina and Anglo women, but it appears to be a greater risk factor for U.S. born Latinas, as they have higher mortality from diabetes. Among Latinas, diabetes ranks as the third leading cause of death.

DESIGN NARRATIVE:

Hispanic Americans, in particular postmenopausal Hispanic women, have an increased prevalence of type 2 diabetes, and a greater incidence of diabetes complications than non-Hispanic whites. The LLP will comprehensively evaluate a multiple risk factor intervention (diet, physical activity, stress management, social support, and smoking cessation) in a randomized effectiveness trial that will be offered in English and Spanish. The research team has shown that a similar theory-based comprehensive program, Mediterranean Lifestyle Program (MLP), is effective in improving behavioral, psychosocial, quality of life, and physiologic outcomes in postmenopausal Anglo women with type 2 diabetes. Though the results are promising, four important research issues must be addressed before such a program is ready to be put into practice. This study focuses on the following questions: 1) How should the structure and content of the MLP be modified to address the cultural characteristics of Latinas?; 2) Will the program succeed if offered within a large health plan that serves minority populations (i.e., the Kaiser Permanente site in Denver, CO)?; and 3) What are the economic implications of the LLP? The Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) evaluation framework will be used to assess how the program impacts certain dimensions that are important for carry over into clinical practice. Primary outcomes of this study will include change in behavioral measures. Secondary outcomes will include impacts on quality of life, physiologic measures, member satisfaction, and cost-effectiveness. The investigators will also study the relationship between cultural variables in this Hispanic population (e.g., family and social support; group cohesion; and acculturation) and program participation and outcomes. Substantial impacts of this study on public health include: 1) intervening with a high-risk, underserved population; 2) focusing on multiple critically important lifestyle behaviors known to reduce risk for CHD; 3) testing maintenance of behavioral changes; 4) employing methodology to estimate the program's readiness to be put into practice; and (5) measuring the robustness, reach, and cost-effectiveness of the program.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Postmenopausal
* Latina

Exclusion criteria:

* Cognitive impairment or inability to comprehend program
* Has other life-threatening illnesses
* Planning to move from the area during the study

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2006-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean Diet, physical activity, stress management, and smoking cessation protocols | Measured at baseline, 6, 12, and 24 months
Hemoglobin A1c | Measured at baseline, 6, 12, and 24 months

SECONDARY OUTCOMES:
Social support | Measured at baseline, 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Toobert, PhD, Study Chair — Oregon Research Institute
Locations (1):
- Institute for Health Research, Denver, Colorado, United States

REFERENCES:
- [Derived] Toobert DJ, Strycker LA, King DK, Barrera M Jr, Osuna D, Glasgow RE. Long-term outcomes from a multiple-risk-factor diabetes trial for Latinas: inverted exclamation markViva Bien! Transl Behav Med. 2011 Sep;1(3):416-426. doi: 10.1007/s13142-010-0011-1. PMID 22022345
- [Derived] Toobert DJ, Strycker LA, Glasgow RE, Osuna D, Doty AT, Barrera M, Geno CR, Ritzwoller DP. Viva bien!: Overcoming recruitment challenges in a multiple-risk-factor diabetes trial. Am J Health Behav. 2010 Jul-Aug;34(4):432-41. doi: 10.5993/ajhb.34.4.5. PMID 20218755
- [Derived] Osuna D, Barrera M Jr, Strycker LA, Toobert DJ, Glasgow RE, Geno CR, Almeida F, Perdomo M, King D, Doty AT. Methods for the cultural adaptation of a diabetes lifestyle intervention for Latinas: an illustrative project. Health Promot Pract. 2011 May;12(3):341-8. doi: 10.1177/1524839909343279. Epub 2009 Oct 20. PMID 19843703